CLINICAL TRIAL: NCT07362251
Title: Evaluation of the Acceptability of a Multi-strain Probiotic Supplement (Smile Probio 45B) in Healthy Adults: an Open-label Pilot Study
Brief Title: Evaluation of the Acceptability of a Multi-strain Probiotic Supplement (Smile Probio 45B) in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Vaios Svolos, Dietitian, Postdoctoral Researcher, University of Thessaly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25 / 28.03.2025
Record Dates: First submitted 2025-12-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: acceptability; probiotic; multi strain
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic Intervention (Experimental): Participants will receive probiotic supplement for 4 weeks
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Participants will receive probiotic supplement: 1 capsule daily for 2 weeks, followed by 3 capsules daily for 2 weeks.

SUMMARY:
The goal of this clinical trial is to examine the compliance and acceptability of the probiotic Smile Probio 45B in healthy adults, as well as its effect on gastrointestinal symptoms, fatigue levels, and quality of life.

Specifically, the study examines the effect of probiotic intake on improving health-related quality of life, reducing self-reported gastrointestinal symptoms such as bloating, as well as regulating stool consistency and frequency. In addition, its impact on participants' self-reported energy levels is investigated, with a particular emphasis on reducing fatigue symptoms.

Participants will:

* take 1 capsule daily (with a main meal) during the first and second week of the intervention, and 3 capsules daily (after each main meal) during the third and fourth week of the intervention, for a total duration of 30 days.
* complete a three-day food record on a weekly basis.
* record their daily bowel habits, including the number of bowel movements and their consistency/form, according to the Bristol Stool Chart, which will be provided to them.
* complete questionnaires assessing health-related quality of life [WHOQOL-BREF (World Health Organization Quality of Life)],a health status questionnaire [EQ-5D (EuroQol-5D)] and a questionnaire evaluating energy levels and fatigue [Chalder Fatigue Scale (CFQ)].
* complete, at baseline and at the end of each intervention week a weekly symptom assessment questionnaire.
* undergo body composition assessment at the beginning, midpoint, and end of the study.
* complete an acceptability questionnaire at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Body Mass Index (BMI) >18 kg/m² and <30 kg/m²
* No use of antibiotics in the past month
* Willingness to provide informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Age under 18 years
* Diagnosis of a chronic autoimmune disease (e.g., Crohn's disease, ulcerative colitis, rheumatoid arthritis, psoriasis)
* Diagnosis of type I or II diabetes
* Current use of immunosuppressive medications
* Current use of antibiotics or use of antibiotics within the past month
* Current use of other supplements such as probiotics, prebiotics, or synbiotics
* Kidney or liver disease
* Self-reported allergy to any component of the probiotic
* Psychological conditions affecting the ability to provide informed consent (e.g., dementia, psychosis, substance use)
* Gastrointestinal surgery within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Daily compliance and stool consistency using the Bristol Stool Form Scale | From enrollment to the end of treatment at 4 weeks
  Participants will record their daily compliance and stool consistency using the Bristol Stool Form Scale. Adherence to the intervention will be evaluated by recording the number of days the probiotic was consumed. To prevent potential non-compliance, participants weill be contacted via telephone on a weekly basis. At the conclusion of the study, participants will be asked to return all empty packaging and any remaining capsules.
Acceptability of the probiotic using an acceptability questionnaire | Immediately after the intervention
  At the end of the intervention, participants will complete an acceptability questionnaire, including questions regarding ease of use of the probiotic, perceived product safety, and intention to recommend it to others.

SECONDARY OUTCOMES:
Effect of Smile Probio 45B on gastrointestinal symptoms | From enrollment to the end of treatment at 4 weeks
  Participants will complete a weekly symptom assessment questionnaire at baseline and at the end of each week of the intervention. The questionnaire will include questions on how frequently they experienced skin reactions, headaches, changes in bowel movement frequency, nausea, diarrhea, constipation, abdominal bloating, abdominal pain, flatulence, acidic taste, and sleep difficulties. Responses will be recorded on a Likert scale (not at all = 1, rarely = 2, occasionally = 3, often = 4, and daily = 5). Higher scores mean a worse outcome.
Effect of Smile Probio 45B on fatigue levels | From enrollment to the end of treatment at 4 weeks
  Fatigue levels will be assessed using the Chalder Fatigue Scale (CFS), which consists of 11 Likert-scale questions designed to distinguish between physical and mental fatigue. Responses will be scored using the Likert method (0-3), yielding a total fatigue score ranging from 0 to 33, with higher scores indicating greater fatigue severity.
  Permission for the use of this questionnaire was requested and obtained from the respective creator.
Effect of Smile Probio 45B on quality of life using the EQ-5D-5L questionnaire | From enrollment to the end of treatment at 4 weeks
  Quality of life (QoL) will be assessed using EQ-5D-5L, a standardized instrument for measuring generic health status, comprising five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a Visual Analogue Scale (VAS). The EQ-5D-5L index score will be calculated using the validated country-specific value set, converting health states into a single index value ranging from 0 to 1, where higher values indicate better health-related quality of life.
Effect of Smile Probio 45B on quality of life using the WHOQOL-BREF questionnaire | From enrollment to the end of treatment at 4 weeks
  Quality of life (QoL) will be assessed using the WHOQOL-BREF (World Health Organization Quality of Life-Abbreviated version), which consists of 26 items rated on a 5-point Likert scale and evaluates four domains: physical health, psychological health, social relationships, and environment, along with two items assessing overall quality of life and general health. Domain scores will be calculated and transformed to a 0-100 scale according to World Health Organization guidelines, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Education, Sport Science and Dietetics, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No